CLINICAL TRIAL: NCT03975257
Title: Application of Ectoin Lozenges (EHT02) in Patients With Oropharyngeal Allergic Symptoms
Brief Title: Ectoin Lozenges (EHT02) in the Treatment of Oropharyngeal Allergic Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: btph-021-2018-EHT02
Record Dates: First submitted 2019-01-22; First posted 2019-06-05 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preventive application of EHT02 (Experimental): application of one Ectoin Lozenge before SLIT-initiation
  Interventions: Device: Medical Device: Ectoin Lozenge
- Therapeutic application of EHT02 (Experimental): application of one Ectoine Lozenge after SLIT-initiation
  Interventions: Device: Medical Device: Ectoin Lozenge
- No application of EHT02 (No Intervention): SLIT-Initiation without Ectoin Lozenge

INTERVENTIONS:
Device: Medical Device: Ectoin Lozenge — Application of Ectoin Lozenge (EHT02) in accordance with the instructions for use
  Other Names: EHT02
  Arms: Preventive application of EHT02; Therapeutic application of EHT02

SUMMARY:
The goal of this multicentric, prospective, randomised, controlled study (§23b German Act on Medical Devices (MPG)) is to investigate the efficacy of Ectoin Lozenges (EHT02) in treatment and prevention of oropharyngeal allergic symptoms.

DETAILED DESCRIPTION:
The immune system of humans can show an overreaction to proteins from the environment (allergic reaction). Triggers of these allergic reactions may be e.g. pollen, dust mites, mold or animal hair. Common allergic symptoms include itchy, stuffy, runny nose, sneezing, itchy and watery eyes and respiratory complaints. Allergen-specific immunotherapy is the only treatment that eliminates the causes of allergic disease. An example of such immunotherapies is the sublingual immunotherapy (SLIT). During SLIT, side effects may occur such as local oropharyngeal reactions, e.g. manifesting as itching, swelling or irritation.

The current study aims to investigate the efficacy of Ectoin Lozenges (EHT02) in patients suffering from oropharyngeal allergic symptoms. The symptoms are induced by SLIT.

Patients are dedicated to one of three groups: a) preventive application of Ectoin Lozenges before SLIT-initiation, b) therapeutic application of Ectoin Lozenges after SLIT-initiation or c) control: SLIT-initiation without application of Ectoin Lozenges.

The symptoms itching, swelling and irritation of mouth, lips and throat will be documented by the patients once 30 minutes after SLIT-initiation.

ELIGIBILITY:
Inclusion criteria:

* initiation of a SLIT
* minimum age of 18 years
* written consent of the patient

Exclusion criteria:

* Surgical Procedures in the mouth and throat region prior to the study
* patients with known intolerance to one of the substances used
* pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
cumulative score of allergic symptoms of the lips evaluated by the patient | about 30 minutes after SLIT-initiation
  about 30 minutes after SLIT-initiation patients will assess allergic symptoms of the lips (swelling, itching and irritation) on a 4 point scale (0=none to 3=severe)
cumulative score of allergic symptoms of the mouth evaluated by the patient | about 30 minutes after SLIT-initiation
  about 30 minutes after SLIT-initiation patients will assess allergic symptoms of the mouth (swelling, itching and irritation) on a 4 point scale (0=none to 3=severe)
cumulative score of allergic symptoms of the throat evaluated by the patient | about 30 minutes after SLIT-initiation
  about 30 minutes after SLIT-initiation patients will assess allergic symptoms of the throat (swelling, itching and irritation) on a 4 point scale (0=none to 3=severe)

SECONDARY OUTCOMES:
Incidence of adverse events/serious adverse events | through study visit (participation encompasses 1 visit of approx. 60 min duration)
  All occurring adverse events/serious adverse events will be documented during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bilstein, Dr., Study Director — CSO
Locations (8):
- Germany (8):
  - Facharzt f. HNO-Heilkunde, Aachen
  - Fachärztin für Hals-Nasen-Ohrenheilkunde, Bad Schönborn
  - Facharzt f. Dermatologie ruhrDerm GbR, Bochum
  - Facharzt für Lungen- und Bronchialheilkunde, Bonn
  - Facharzt für Haut und Geschlechtskrankheiten, Gelsenkirchen
  - Arzt für Hals-Nasen-Ohrenheilkunde, Allergologie, Umweltmedizin, Naturheilverfahren, Flugmedizin, Taucherarzt (GTÜM), Heidelberg
  - Fachärztin f. HNO-Heilkunde, Allergologie, Jülich
  - Facharzt für Hals-Nasen-Ohrenheilkunde, Allergo GmbH Stuttgart, Klinische Prüfstelle Schorndorf, Schorndorf